CLINICAL TRIAL: NCT06022900
Title: The Impact of Two Distinct Health Education Approaches on Mammography Self-Efficacy, Health Beliefs, and Screening Program Participation: a Randomized Controlled Trial
Brief Title: The Effect of Health Education on Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, PhD RN, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BREASTCANCER
Record Dates: First submitted 2023-08-21; First posted 2023-09-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Mammography; Health Education; Online Education; Home Visit
MeSH Terms: conditions — Breast Neoplasms; Health Education

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomised control trial
Who Masked: Participant
Masking Description: Single (Participant); single blind study, participants do not know their group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): During the study period, this group participated in the standard breast cancer screening program, which is a nationwide health initiative implemented throughout the country to promote early detection and prevention of breast cancer.
- Online training group (Experimental): Alongside the standard breast cancer screening services, participants in this group were offered comprehensive online health education that emphasized both breast cancer awareness and prevention strategies. Additionally, they received a digital educational brochure designed to enhance their understanding of the disease. Four weeks after their enrollment in the study, participants were contacted via phone to reinforce the significance of regular screenings and to provide them with a summary of essential information regarding the benefits of early detection.
  Interventions: Behavioral: Online training group
- Face-to-face training group (Experimental): In addition to the standard breast cancer screening services, individuals in this group received tailored in-person health education regarding breast cancer and its prevention through comprehensive home visits, which included a well-designed training brochure. At the conclusion of the fourth week following their enrollment in the study, participants were contacted via phone to emphasize the critical importance of regular screening. During this call, they were provided with a concise summary of key information aimed at reinforcing the benefits of early detection and encouraging ongoing participation in screening programs.
  Interventions: Behavioral: Face-to-face training group

INTERVENTIONS:
Behavioral: Online training group — online health education with video call
  Arms: Online training group
Behavioral: Face-to-face training group — Face-to-face health education with home visit
  Arms: Face-to-face training group

SUMMARY:
Objective: This study aimed to explore how face-to-face and online health education influenced several factors related to breast cancer, including individuals' self-reported knowledge of breast cancer and mammography, perceptions of the benefits and barriers to mammography, self-confidence in undergoing mammography, and the rates of participation in screening programs.

Materials and Methods: This research utilized a parallel group design within a single-blind randomized controlled trial framework. A total of 126 healthy participants were recruited, equally divided into three groups of 42, from individuals enrolled at the Toprakkale Family Health Center between January and July 2023, all of whom met the eligibility requirements.In this study, a 10-point Visual Analogue Scale, along with the mammography benefit and barrier perception sub-dimensions from Champion's Health Belief Model Scale and the Mammography Self-Efficacy Scale, were utilized for participants to self-assess their knowledge regarding breast cancer and mammography. While the control group received standard care, the face-to-face education group benefited from health education and informational brochures delivered through home visits, supplemented by a follow-up reminder call. Meanwhile, the online training group received health education and digital brochures via video calls, along with one reminder session. Following a two-month follow-up period, data from the three groups were compared using One-Way Analysis of Variance and the Kruskal-Wallis H test. Multiple comparisons were conducted using Tukey's test and Dunn's test, while Generalized Linear Models were employed for assessing group and time differences.

DETAILED DESCRIPTION:
This investigation was structured as a single-blind, parallel-group randomized controlled trial, taking place at the Toprakkale Family Health Center in Osmaniye Province from January to July 2023. A power analysis indicated that at least 96 participants were necessary to achieve a significant effect size (d=0.18) with a 95% power and a 0.05 error margin. The G Power 3.1.9.2 software facilitated these calculations. To mitigate the potential impact of data loss, an additional 30% of participants were included, resulting in a final sample size of 126 individuals, with each of the three groups consisting of 42 participants.

Women aged 40 to 69 who visited the Family Health Center were informed about the study's objectives and subsequently invited to participate. After obtaining consent, the volunteers were screened against the established inclusion criteria. The researchers provided detailed information about the study's goals and handed out Form I to those deemed eligible.

For the purpose of randomization, a block randomization technique was employed, assigning participants to groups based on their order of arrival at the center according to the pre-established randomization list. The control group did not receive any intervention during the study duration. Participants in the online training group were offered digital health education along with an electronic brochure, while those in the face-to-face training group received personalized health education through home visits and a physical training brochure.

Four weeks into the intervention, both the online and face-to-face groups received reminder calls to encourage ongoing engagement. At the conclusion of the eight-week period, all participants completed Form II, allowing for the evaluation of outcomes across all groups.

ELIGIBILITY:
Inclusion Criteria:

Must voluntarily agree to participate in the research. Must be literate in Turkish. Must be aged between 40 and 69 years. Must identify as a woman. Must have access to the necessary technology for video calls.

Exclusion Criteria:

Any barriers to effective communication. Currently pregnant or in the postpartum period. Currently breastfeeding. Having undergone a mammogram within the past two years. A history of benign breast disease or breast cancer. A family history of breast cancer.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — intervention for breast cancer
Enrollment: 126 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy Scale for Mammography | 60 days
  The scale comprises 10 items, each rated on a 5-point Likert type format. The total score that can be achieved ranges from 10 to 50.

SECONDARY OUTCOMES:
Champion's Health Belief Model Scale | 60 days
  Description: This study focused on two specific sub-dimensions of the scale: the perception of benefits associated with mammography and the perception of barriers to mammography. The benefits sub-dimension comprises five items, while the barriers sub-dimension includes eleven items. In this scale, the perceived benefits of mammography are scored on a scale from 5 to 25 points, whereas the perceived barriers to mammography are scored from 11 to 55 points.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Ozdemir, PhD, Principal Investigator — Sağlık Bilimleri Üniversitesi Gülhane Hemşirelik Fakültesi
Locations (1):
- University of Health Sciences, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No